CLINICAL TRIAL: NCT04075331
Title: A Randomised Controlled Trial of Mepolizumab Initiated Following Admission to Hospital for a Severe Exacerbation of Eosinophilic COPD
Brief Title: Mepolizumab for COPD Hospital Eosinophilic Admissions Pragmatic Trial
Acronym: COPD-HELP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0690
Record Dates: First submitted 2019-05-23; First posted 2019-08-30 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2023-11

CONDITIONS: COPD; Eosinophilia
Keywords: COPD; eosinophilia; Chronic Obstructive Pulmonary Disorder; Mepolizumab
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Eosinophilia | interventions — mepolizumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mepolizumab (Experimental): Mepolizumab
  Interventions: Drug: Mepolizumab
- Placebo (Placebo Comparator): Saline solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mepolizumab — Mepolizumab 100mg subcutaneous injection
  Arms: Mepolizumab
Drug: Placebo — Saline solution for subcutaneous injection
  Other Names: Saline solution
  Arms: Placebo

SUMMARY:
This is a single-centre, double-blinded, randomised, placebo controlled trial comparing mepolizumab 100mg versus placebo in patients with eosinophilic COPD, started following their index admission to hospital.

DETAILED DESCRIPTION:
Patients admitted to hospital with an exacerbation of COPD are at high risk of readmission, of which a proportion are driven by eosinophilic inflammation. Whilst oral corticosteroids are beneficial in exacerbations, a considerable proportion of patients experience treatment failure, with 50% of patients readmitted within 3 months (www.RCPLondon.ac.uk).

Therapy, such as mepolizumab, reduces eosinophil count and has been shown to reduce exacerbation frequency when given in the stable state in both eosinophilic asthma (Papi et al. 2018) and COPD (Yousef, in press).

The investigators hypothesise that starting mepolizumab at the time of a hospitalisation for an exacerbation of COPD in patients with significant eosinophilia will result in a reduction in readmission to hospital in a high risk population.

Therefore, 238 participants will be recruited over an 18-month period and will be randomised into a 48-week treatment period in which they will receive monthly subcutaneous injections of either 100 mg mepolizumab or placebo. Secondary outcomes will be measured at baseline (week 0), 4 weeks, 8 weeks, 12 weeks, 24 weeks, 36 weeks and 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms typical of COPD when stable (baseline eMRC dyspnoea grade 2 or more).
2. A clinician defined exacerbation of COPD requiring admission to hospital.
3. Serum eosinophil count of ≥ 300 cells/μL either at time of admission or at any one time in the preceding 12 months.
4. Smoking pack years ≥10 years.
5. Age ≥ 40 years.
6. Established on inhaled corticosteroids (ICS) prior to this admission.
7. Willing and able to consent to participate in trial.
8. Able to understand written and spoken English.

Exclusion Criteria:

1. COPD patients without eosinophilia (defined as persistently < 300 cells/μL within the last 12 months).
2. Other conditions that may be the cause of eosinophilia (such as hypereosinophilic syndrome, eosinophilic granulomatosis, eosinophilic oesophagitis or parasitic infection).
3. Patients whose treatment is considered palliative (life expectancy < 6 months).
4. Other respiratory conditions including active lung cancer, interstitial lung disease, primary pulmonary hypertension or any other conditions that in the view of the investigator will affect the trial.
5. Known history of anaphylaxis or hypersensitivity to mepolizumab or any of the excipients (sucrose, sodium phosphate dibasic heptahydrate, polysorbate 80).
6. Unstable or life-threatening cardiac disease including myocardial infarction or unstable angina in the last 6 months, unstable or life-threatening cardiac arrhythmia requiring intervention in the last 3 months and New York Heart Association (NYHA) Class IV heart failure.
7. Decompensated liver disease or cirrhosis.
8. Pregnant, breastfeeding, or lactating women. Women of child-bearing potential must agree to use appropriate methods of birth control and have a negative blood serum pregnancy test performed after randomisation but prior to first dosing with randomised treatment.*
9. Participation in an interventional clinical trial within 3 months of visit 1 or receipt of any investigational medicinal product within 3 months or 5 half-lives.
10. Known blood born infection (e.g. HIV, hepatitis B or C).

    * Women of child bearing potential (WOCBP) - A woman is defined as being of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal, unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Time from randomisation to next hospital readmission or death (all cause) | 48 weeks
  To evaluate the efficacy of mepolizumab initiated following hospitalisation on future hospital readmission or death (all cause) compared with placebo and standard medical therapy in severe exacerbations of eosinophilic COPD.

SECONDARY OUTCOMES:
Time from randomisation to first hospital readmission or death due to a respiratory cause | 48 weeks
Total number of hospital readmissions all cause over 48 weeks | 48 weeks
  (adjusted for time minimum 24 weeks of trial treatment)
Total number of moderate exacerbations over 48 weeks | 48 weeks
  (adjusted for time minimum 24 weeks of trial treatment)
Time from randomisation to treatment failure | 48 weeks
  (defined as readmission, need for further treatment or death)
Time from randomisation to death (all cause) | 48 weeks
Time from randomisation to death (respiratory cause) | 48 weeks
Time from randomisation to first hospital readmission (all cause) | 48 weeks
Time from randomisation to first hospital readmission (respiratory cause) | 48 weeks
Length of index hospital admission | 48 weeks
  Time from admission to discharge of first hospital admission
Extended Medical Research Council dyspnoea score (eMRC) | Weeks 0, 4, 8, 12, 24, 36, 48
  This scale measures perceived respiratory disability. Participants rate their grades of breathlessness on a scale of 1 (least) to 5 (worst). The extension divides the grade 5 rating into 'a' (independent) and 'b' (dependent) to establish dependence on others for washing and dressing.
St George's Respiratory Questionnaire (SGRQ) | Weeks 0, 4, 8, 12, 24, 36, 48
  This 50-item questionnaire measures health status (quality of life) in patients with diseases of airway obstruction. Scores are broken down into 'symptoms' (normal participant range 9-15), 'activity' (normal participant range 7-12), 'impacts' (normal participant range 1-3), and a total score (normal participant range 5-7). Higher scores indicate poorer health status.
COPD Assessment Tool (CAT) | Weeks 0, 4, 8, 12, 24, 36, 48
  The COPD Assessment Test (CAT) is a questionnaire for people with Chronic Obstructive Pulmonary Disease (COPD). It is designed to measure the impact of COPD on a person's life, and how this changes over time. Scores range from 0-40, with higher scores indicating greater impact of COPD on a patient's life.
Warwick-Edinburgh Mental wellbeing scale (WEMWBS) | Weeks 0, 4, 8, 12, 24, 36, 48
  This scale measures mental wellbeing using a 14-item scale. The scoring range for each item is from 1 - 5 and the total score is from 14-70, with higher scores indicating better mental wellbeing.
London Chest Activities of Daily Living Questionnaire (LCADL) | Weeks 0, 4, 8, 12, 24, 36, 48
  This 15-item questionnaire measures dyspnoea during routine daily activities in patients with COPD. It consists of four components: 'Self-care', 'Domestic', 'Physical' and 'Leisure'. Patients score from 0: 'I wouldn't do anyway', to 5: 'Someone else does this for me (or helps)', with higher scores representing maximal disability.
Short physical performance battery (SPPB) | Weeks 0, 4, 8, 12, 24, 36, 48
  This assessment measures lower extremity functioning in older individuals. Lower scores indicate greater impairment.
Physical activity using accelerometry | Weeks 0, 4, 8, 12, 24, 36, 48
Handgrip Strength | Weeks 0, 4, 8, 12, 24, 36, 48
Total Serum eosinophil count (inflammatory markers) | Weeks 0, 4, 8, 12, 24, 36, 48
Percentage sputum eosinophil count (inflammatory markers) | Weeks 0, 4, 8, 12, 24, 36, 48
Adverse Events (AEs) | 48 weeks
Serious Adverse Events (SAEs) | 48 weeks
Heart Rate (beats per minute) | Weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48
Blood pressure (systolic/diastolic mmHg) | Weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48
Temperature (degrees) | Weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Brightling, Study Chair — University of Leicester; Neil Greening, Principal Investigator — University of Leicester
Locations (1):
- NIHR Biomedical Research Centre, Respiratory, Leicester, Leicestershire, United Kingdom

REFERENCES:
- [Derived] Flynn CA, McAuley HJC, Elneima O, Aung HWW, Ibrahim W, Ward TJC, Bourne M, Thornton TD, Mistry V, Gilbert HR, Waheed G, Wright AKA, Evans RA, Steiner MC, Brookes CL, Brightling CE, Greening NJ. Mepolizumab for COPD with Eosinophilic Phenotype following Hospitalization. NEJM Evid. 2025 Jun;4(6):EVIDoa2500012. doi: 10.1056/EVIDoa2500012. Epub 2025 Apr 30. PMID 40305842